CLINICAL TRIAL: NCT03220295
Title: Study of the M1 Positive Allosteric Modulator VU0467319
Brief Title: Putative Cognitive Enhancer VU319
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Paul Newhouse, MD/PI, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VU319
Record Dates: First submitted 2017-07-06; First posted 2017-07-18 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind safety study. The pharmacist is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Dose Escalation of VU319 - Dose 1 (Experimental): Dose Escalation of VU319
  Interventions: Drug: Dose Escalation of VU319
- Placebo - Dose 1 (Placebo Comparator): Dose Escalation of Placebo
  Interventions: Drug: Placebo Dose Escalation
- Single Dose of VU319 under Fed State (Experimental): Single dose of VU319 (50% of the maximum tolerated dose) 30 minutes after a High Fat Standard Breakfast
  Interventions: Drug: Single Dose of VU319; Other: Fed State
- Single Dose of Placebo under Fed State (Placebo Comparator): Single dose of Placebo 30 minutes after a High Fat Standard Breakfast
  Interventions: Drug: Single Dose Placebo; Other: Fed State
- Single Dose of VU319 under Fasted State (Experimental): Single dose of VU319 (50% of the maximum tolerated dose) after overnight fast
  Interventions: Drug: Single Dose of VU319; Other: Fasted State
- Single Dose of Placebo under Fasted State (Placebo Comparator): Single dose of placebo after overnight fast
  Interventions: Drug: Single Dose Placebo; Other: Fasted State
- Dose Escalation of VU319 - Dose 2 (Experimental): Dose Escalation of VU319
  Interventions: Drug: Dose Escalation of VU319
- Dose Escalation of VU319 - Dose 3 (Experimental): Dose Escalation of VU319
  Interventions: Drug: Dose Escalation of VU319
- Dose Escalation of VU319 - Dose 4 (Experimental): Dose Escalation of VU319
  Interventions: Drug: Dose Escalation of VU319
- Dose Escalation of VU319 - Dose 5 (Experimental): Dose Escalation of VU319
  Interventions: Drug: Dose Escalation of VU319
- Placebo - Dose 2 (Placebo Comparator): Dose Escalation of Placebo
  Interventions: Drug: Placebo Dose Escalation
- Placebo - Dose 3 (Placebo Comparator): Dose Escalation of Placebo
  Interventions: Drug: Placebo Dose Escalation
- Placebo - Dose 4 (Placebo Comparator): Dose Escalation of Placebo
  Interventions: Drug: Placebo Dose Escalation
- Placebo - Dose 5 (Placebo Comparator): Dose Escalation of Placebo
  Interventions: Drug: Placebo Dose Escalation

INTERVENTIONS:
Drug: Single Dose of VU319 — Single dose of VU319
  Arms: Single Dose of VU319 under Fasted State; Single Dose of VU319 under Fed State
Drug: Single Dose Placebo — Single dose of placebo
  Arms: Single Dose of Placebo under Fasted State; Single Dose of Placebo under Fed State
Other: Fed State — drug is given 30 minutes after a high fat breakfast
  Arms: Single Dose of Placebo under Fed State; Single Dose of VU319 under Fed State
Other: Fasted State — drug is given after an overnight fast
  Arms: Single Dose of Placebo under Fasted State; Single Dose of VU319 under Fasted State
Drug: Dose Escalation of VU319 — dose levels of the cohorts will be increased step wise
  Arms: Dose Escalation of VU319 - Dose 1; Dose Escalation of VU319 - Dose 2; Dose Escalation of VU319 - Dose 3; Dose Escalation of VU319 - Dose 4; Dose Escalation of VU319 - Dose 5
Drug: Placebo Dose Escalation — dose levels of the cohorts will be increased step wise
  Arms: Placebo - Dose 1; Placebo - Dose 2; Placebo - Dose 3; Placebo - Dose 4; Placebo - Dose 5

SUMMARY:
This is a safety study of the molecule VU319 to ascertain pharmacokinetic and pharmacodynamic data and test cognitive enhancement in healthy volunteers.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is a chronic and irreversible neurodegenerative disease characterized by the deterioration of memory and other cognitive functions, progressive impairments in normal daily living, and severe neuropsychiatric symptoms and behavioral disturbances1,2. Currently, there is no available prevention or cure for AD. Therapeutic strategies for the cognitive impairments in AD involve only symptomatic treatments, primarily through enhancement of cholinergic neurotransmission using AChEIs1,2.

This first trial will be First-in-Human single ascending dose (SAD) phase 1 trial in healthy volunteers. One dose will be selected for expansion and evaluation of the effect of food on bioavailability. This Phase I trial, if successful, would serve as the basis for the design of multiple ascending dose (MAD) Phase I trial.

Primary objectives To establish the safety and tolerability of single dose (up to VU319 steady state) VU319 administration in healthy volunteers To establish the maximum tolerated dose of single dose (up to VU319 steady state) VU319 administration in healthy volunteers To characterize the plasma pharmacokinetics and urinary excretion of VU319 and metabolite after single dose oral administration in healthy volunteers Secondary objectives To establish the effect of food on the bioavailability and pharmacokinetic parameters of VU319 in healthy volunteers Exploratory Objectives To gain preliminary evidence that tolerable doses of VU319 engage central M1 receptors by 1) altering/enhancing cognitive performance, and 2) enhancing cortical event related potentials (ERP) as a measure of increased cognitive function in healthy volunteers This will be a double blind, randomized, placebo controlled, and sequential dose escalation in male or female healthy volunteers. Gender will be balanced to the extent possible. Volunteers will receive oral VU319 single dose administration in the fasted state. Subjects meeting entry criteria will be enrolled in successive dose escalating cohorts of 8 subjects each (2 placebo and 6 active drug per dose level). The dose levels will be tested sequentially until the Maximum Tolerated Dose (MTD) is reached, or saturation of exposure occurs, or sustained VU319 plasma level above the safe daily exposure determined from animal toxicokinetic studies is achieved.

The food effect sequence will be double blind, placebo controlled, two sequences, balanced and sequential cross-over in 12 healthy male or female volunteers (2 placebo and 10 active drug). Volunteers will receive oral VU319 single dose administration repeated once under either the fed (i.e. high fatty meal per FDA recommendations) or fasted state. The order of the two periods will be randomized and balanced with 6 subjects receiving treatment in the fed/fast or fast/fed order, respectively.

Clinical safety endpoints include adverse event and symptoms data, vital signs (HR, BP, Respiratory Rate, body weight), 12-lead ECG changes, and laboratory safety assessments (hematology, plasma biochemistry, coagulation, urinalysis).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 through 55 years, inclusive.
* Body mass index 18 through 32 kg/m2
* Determined as healthy based on screening medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG (QTc interval with Fridericia's correction method recorded on screening and predose must be less than 450 msec for male and less than 470 in females).
* Clinical laboratory test result without clinically significant abnormalities at screening and at admission.
* Negative tests for Hepatitis B surface antigen, hepatitis C virus antibodies and human immunodeficiency virus (HIV-1 or HIV-2) antibody at screening.
* Nonsmokers (use of any nicotine containing product) or ex-smokers (have ceased smoking for at least 6 months and do not use any drug for smoking cessation).
* Negative screen for alcohol and drugs of abuse at screening and admission.
* For Women: Must have no child-bearing potential by reason of surgery or at least 1 year post-menopausal (i.e. 12 months without menstrual period), or menopause confirmed with an estradiol level of < 30 pg/mL and follicle-stimulating hormone level of > 40 IU/L at screening.
* For Men: Must be infertile (at least 3-months post-vasectomy), or truly abstinent of heterosexual intercourse, or heterosexual partner is not of child-bearing potential, or must agree to use an effective method of contraception (condom or occlusive cap with spermicidal foam/gel/film/cream/suppository) through the study and for 28 days after last dose of study drug.
* Able and willing to be available for the duration of the study.
* Willing and able to give written informed consent to participate.
* Able to understand and comply with protocol instructions.
* Agrees not to receive any vaccination within 21 days prior to admission and through Day 7 after final discharge.
* Agrees not to use nonprescription drugs, including vitamins, antacids, and herbal and dietary supplements within 7 days prior to admission and through 7 days after final discharge. Acetaminophen may be used at doses of ≤ 1 g/day, and ibuprofen may be used at doses of ≤ 1.2 g/day starting no earlier than 48 hours after discharge.
* Agrees not to use nicotine-containing products from screening through 48 hours after discharge.
* Agrees not to consume alcohol for the 72 hours prior to admission and through 48 hours after discharge.
* Agrees not to eat grapefruit or drink grapefruit juice within 7 days prior to admission and through 24 hours after discharge.
* Agrees to not drink caffeinated drinks from 72 hours prior to admission to discharge.
* Agrees not to eat or drink (except water) for 8 hours before and 4 hour after dosing for all SAD cohort participants (applicable to the Food Effect Cohort participants only for the fasted dose).
* Agrees to eat the high-fat standard breakfast 30 minutes pre-dose for participants in Food Effect Cohort.

Exclusion Criteria:

* Individuals with significant previous or ongoing disease or disorder, on the basis of history, physical exam, ECG, and laboratory tests, including for example: Cardiovascular diseases; hypertension; cancer or neoplasia; diabetes; hepatic, endocrine, metabolic, respiratory, renal, gastrointestinal (except appendectomy), dermatological or hematological disorders, Axis I or II psychiatric, substance use, or cognitive disorders.
* Clinically significant infection or inflammation at time of screening or admission.
* Clinically significant abnormalities upon physical/neurological exam at screening.
* Acute gastrointestinal symptoms (e.g. nausea, vomiting, diarrhea) at time of screening or admission
* History of seeking advice from a physician or counselor for abuse or misuse of alcohol, non-medical drugs, medicinal drugs or other substance abuse, for example, solvents.
* Any current or previous use of Class A drugs such as illicit opiate use, cocaine, ecstasy, LSD, and amphetamines (Class B). Volunteers that admit to occasional past use of cannabis will not be excluded as long as they have a negative drugs-of-abuse test at screening and admission and have been abstinent for at least 3 months.
* An alcoholic intake greater than 21 units per week or unwillingness to stop alcohol consumption for the duration of the study. Note: 1 unit = 8 g ethanol (250 mL of beer, 1 glass wine [100 mL], 1 measure spirits [30 mL]).
* Use of medication (including OTC and oral contraceptive agents) within 14 days of admission that may affect the safety of the subject or any study assessment, in the opinion of the investigator.
* Use of prescribed centrally active or psychoactive agents within 28 days from admission.
* Requirement for any medication that would need to be continued during the study.
* Use of any investigational medication within 3 months prior to the start of this study or scheduled to receive an investigational drug during the course of this study.
* Have participated in more than 2 clinical trials within the 12 months prior to screening
* History of blood donation in the last 3 months.
* History of severe allergies or multiple adverse drug reactions.
* Any condition, which compromises ability to give informed consent or to communicate with the investigator as required for the completion of this study.
* The subject has been previously enrolled in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Change in adverse events frequency from Baseline to 144 hours post drug administration
  Frequency of adverse events per ascending dose cohort

SECONDARY OUTCOMES:
Cognitive Battery - Critical Flicker Fusion (CFF) | Baseline, 5 hours post drug administration
  The Critical Flicker Fusion (CFF) task will be used as a test of vigilance. In an ascending trial, the participant presses a button indicating when the frequency of flashing lights, (beginning at 12 Hz and increasing to 50 Hz), has increased to the point that the lights appear to be no longer flashing but rather appear continuously on ("fused"). In a descending trial, beginning at 50 Hz, the participant presses a button when the frequency of apparently fused lights is decreased such that lights begin to appear to be flashing. The participant needs to respond before the frequency hits the upper or lower limit in each trial. The dependent measure is ascending and descending fusion frequency
Cognitive Battery - Choice Reaction Time (CRT) | Baseline, 5 hours post drug administration
  The Choice Reaction Time (CRT) task from the Milford Test Battery will be used. In this task, the subject holds their index finger on a "home" key and monitors an arc of LED lights in front of them. When one of the lights illuminates, the subject lifts their finger from the home key and pushes a key corresponding to the light, thus extinguishing it. The subject then returns their finger to the home key for the next trial. This widely used version of the CRT allows total RT to be broken down into recognition and motor components. The dependent measure are total reaction time (RT), recognition RT, motor RT.
Cognitive Battery - Spatial Selective Attention (Posner Task) | Baseline, 5 hours post drug administration
  A version of the Posner Task of attentional orienting will be used to assess the ability of subjects to disengage attention and shift to a new target. Subjects will be asked to press a button corresponding to the side of the screen on which a stimulus appears. Before the stimulus, a cue will indicate the side on which the stimulus will next appear. This cue will be valid 80% of the time. The validity effect (change in reaction time between valid and invalidity - cued trials).
Cognitive Battery - Continuous Performance Test (Conners) | Baseline, 5 hours post drug administration
  The Conners Continuous Performance Task (CPT). Participants see a string of letters appearing one at a time on a computer screen. Stimuli appear for 300 msec with a response period of 2 sec for a total of 120 trials. Subjects are instructed to press a button whenever a letter appears on the computer screen and they are to not make a response when they see an A followed by an X. The dependent measures are omission and commission errors, hit reaction time, hit RT SE.
Cognitive Battery - Working Memory (N-Back Test) | Baseline, 5 hours post drug administration
  The N-Back Test will be used as a test of verbal working memory. In this task, the subject views a string of consonant letters (except L, W, and Y), one every 3 seconds. Four conditions are presented: 0-back, 1-back, 2-back and 3-back. In each of the 1-back, 2-back, and 3-back conditions, the task is to decide whether the letter currently presented matches the letter that has been presented 1, 2, or 3 back in the sequence. The dependent measures are sensitivity (d') and bias (C) across load conditions (0-3 back).
Cognitive Battery - The Selective Reminding Task (SRT) | Baseline, 5 hours post drug administration
  The Selective Reminding Task (SRT) is a multi-trial verbal list-learning task allowing the examination of acquisition, encoding and retrieval. This standard test has been widely used in studies of cognitive impairment and offers measures of storage into and retrieval from both short term and long-term memory and intrusion errors. In addition to the measures of recall, recall failure, and consistency we add a long-delay (20 min.) recall trial and a recognition trial to assess discrimination and response bias. This task shows excellent predictive validity and test-retest reliability. We have 10 equivalent forms that are balanced for imagery and frequency to insure enough equivalent forms for the multiple repeated administrations necessary in this study. The dependent measures are total (8 trials) word recall and recall failure consistency.
Event-Related Potentials | Baseline, 6 hours post drug administration
  Statistical analysis will focus on a priori selected electrode clusters corresponding to frontal, central, and parietal midline locations (Fz, Cz, Pz in 10-20 notation), which will be confirmed using spatial Principal Components Analysis. Mean amplitudes of the P300 and P600 responses will be calculated within 250-400ms (frontal P3a), 300-500ms (parietal P300), and 500-800ms (parietal P600) temporal windows. These a priori selected windows will also be confirmed using temporal Principal Components Analysis. Repeated measures Analysis of Variance will be used to examine drug-related effects on stimulus processing. The ANOVA design will include Stimulus (2) x Electrode (3) x Test time (2) within-subject factors. To assess the effect of experimental group membership (placebo vs. active) in performance on these tasks, Group (2) will be used as the between-subject factor.
Behavioral Measure - Profile of Mood State (POMS) | Baseline, 4 hours post drug administration
  The Profile of Mood States (POMS) is a relatively new psychological rating scale used to assess transient, distinct mood states. This scale was developed by McNair, Droppleman, and Lorr (1971). Advantages of using this assessment include the simplicity of administration and ease of participant understanding. Another feature of the assessment that is notable is POMS psychological states can be assessed quickly due to the simplicity of the test. POMS can be administered and measured through written or online forums. The POMS measures six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment. A five-point scale ranging from "not at all" to "extremely" is administered by experimenters to patients to assess their mood states.
Behavioral Measure - Brief Psychiatric Rating Scale (BPRS) | Baseline, 1, 3, and 7 hour post drug administration
  Persons having or suspected of having schizophrenia or other psychotic disorder manifest the disorder in multiple ways. The BPRS assesses the level of 24 symptom constructs such as hostility, suspiciousness, hallucination, and grandiosity. It is particularly useful in gauging the efficacy of treatment in patients who have moderate to severe psychoses. It is based on the clinician's observations of the patient's behavior. The rater enters a number for each symptom construct that ranges from 1 (not present) to 7 (extremely severe). The time necessary to complete the interview and scoring can be as little as 20-30 minutes.
Behavioral Measure - Subject Visual Analogue Scale (SVAS) | Baseline, 4 hours post drug administration
  Subject Visual Analog Scales (VAS) will be used consisting of a series of items such as "drowsiness" or "psychomotor agitation" scored on 100 mm lines scored by the subject.
Behavioral Measure - Observer Visual Analogue Scale (SVAS) | Baseline, 1, 3, and 7 hour post drug administration
  Observer Visual Analog Scales (VAS) will be used consisting of a series of items such as "drowsiness" or "psychomotor agitation" scored on 100 mm lines scored by the investigator.
Behavioral Measure - Stanford Sleepiness Scale | Baseline, 14 times over 36 hours post drug administration
  To collect a spectrum of sleepiness indicators across a day, the SSS is administered at two-hour intervals, usually during the waking part of the day. To correlate objective measures and subjective feelings of sleepiness, the SSS may also be administered immediately before and after naps during a multiple sleep latency test.
  The SSS uses the following numeric scale:
  1. Feeling active, vital, alert, and wide awake.
  2. Functioning at a high level but not at peak performance. Able to concentrate.
  3. Relaxed and awake, but not fully alert. Still responsive.
  4. Feeling a little foggy and let down.
  5. Foggy and beginning to lose track of things. Difficult to stay awake.
  6. Sleepy and prefer to lie down. Woozy.
  7. Almost in reverie and cannot stay awake. Sleep onset is imminent.
Behavioral Measure - Physical Symptom Checklist | Baseline, 1, 2, 3, 5, 9 hour after administration
  A checklist of 22 physical symptoms. Each item is rated 1 to 4, with 1 being none and 4 being severe. Total score range from 22 to 88.
Behavioral Measure - Suicide Behaviors Questionnaire (SBQ-R) | Baseline, 4 hours post drug administration
  It consists of four questions. Each of the four questions addresses a specific risk factor: the first concerns presence of suicidal thoughts and attempts, the second concerns frequency of suicidal thoughts, the third concerns the threat level of suicidal attempts, and the fourth concerns likelihood of future suicidal attempts. The first item has often been used on its own in order to assign individuals to a suicidal and a non-suicidal control group for studies. A total score of 7 and higher in the general population and a total score of 8 and higher in patients with psychiatric disorders indicates significant risk of suicidal behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Newhouse, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Poslunsey MS, Wood MR, Han C, Stauffer SR, Panarese JD, Melancon BJ, Engers JL, Dickerson JW, Peng W, Noetzel MJ, Cho HP, Rodriguez AL, Hopkins CR, Morrison R, Crouch RD, Bridges TM, Blobaum AL, Boutaud O, Daniels JS, Kates MJ, Castelhano A, Rook JM, Niswender CM, Jones CK, Conn PJ, Lindsley CW. Discovery of VU0467319: an M1 Positive Allosteric Modulator Candidate That Advanced into Clinical Trials. ACS Chem Neurosci. 2025 Jan 1;16(1):95-107. doi: 10.1021/acschemneuro.4c00769. Epub 2024 Dec 11. PMID 39660766